CLINICAL TRIAL: NCT03968029
Title: Does Wrapping With Bone Marrow Injection Enhance Healing of Meniscal Sutures Into the Non-vascular Area: A Prospective Randomised Study
Brief Title: Does Wrapping With Bone Marrow Injection Enhance Healing of Meniscal Sutures Into the Avascular Area
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Dr. Robin Martin, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MW_OTR
Record Dates: First submitted 2019-05-10; First posted 2019-05-30 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Meniscus Lesion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suturing meniscal augmented (Experimental): Non-vascularised area meniscus tear was sutured and bone marrow was injected under a protective collagen membrane (ChondroGide)
  Interventions: Procedure: suturing meniscal augmented
- Suturing meniscal (Active Comparator): Non-vascularised area meniscus tear was only sutured
  Interventions: Procedure: suturing meniscal

INTERVENTIONS:
Procedure: suturing meniscal augmented — meniscal tear sutured + bone marrow injection/collagen membrane
  Other Names: meniscal wrapping
  Arms: Suturing meniscal augmented
Procedure: suturing meniscal — meniscal tear sutured
  Arms: Suturing meniscal

SUMMARY:
This study will compare meniscal healing of non-vascularised area augmented or not by bone marrow injected under a protective collagen membrane (meniscal wrapping)

DETAILED DESCRIPTION:
Historically, meniscus was considered as none essential for knee joint, and its removal by meniscectomy was the first-line treatment. Many studies have shown a negative progress towards osteoarthritis after meniscus ablation. This approach has gradually changed to preserve this meniscal capital, making way for new treatments as sutures. However the vascular organization of the meniscus is crucial for its cure. The healing potential of lesions in the meniscus non-vascularised aera is considered insufficient, and are often treated by a partial meniscectomy, resulting in a high risk of osteoarthritis. It appears therefore necessary to develop new strategies, as meniscal wrapping, to preserve meniscus presenting this type of damage.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic or traumatic tears of medial or lateral meniscus;
* Tearing affecting: only 2/3 central (= avascular zone) over more than 1 cm OR extending from the peripheral third (= vascularized area) within the avascular zone over more than 1 cm. In this case, preservation of the peripheral third over a width of at least 4 mm from the capsule;
* Single or multiple tears.

Exclusion Criteria:

* Meniscal tears that can not be sutured, reduced / approximated
* Tear creating a meniscal root avulsion
* Partial meniscal tears
* Meniscal tears already sutured
* Cartilage damage in the compartment> grade 2 (ICRS classification)
* Mechanical axis (varus / valgus) ≥ 2 °
* Untreated ligament deficiency
* Osteotomy and / or concomitant ligament reconstruction, with the exception of ACL reconstruction.
* Compromised general health condition (score ASA score> 2)
* BMI ≥30
* Active smoking, drug use
* Allergy to porcine collagen
* Poor compliance

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2017-07-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in integrity and healing of meniscus repair | 12 and 24 months after treatment
  Arthrography (arthro-CT)
Knee injury and Osteoarthritis Outcome Score (KOOS) | baseline and 3, 12 and 24 months after treatment
  Changes in the 5 subscales of KOOS as assessed from baseline to 24 months post-surgery
International Knee Documentation Committee Score (IKDC) | baseline and 3, 12 and 24 months after treatment
  Change in physical pain and function as assessed by IKDC score from baseline to 24 months post-surgery
SF-12 Survey | baseline and 3, 12 and 24 months after treatment
  Change in functional health and well-being as assessed by SF-12 Survey from baseline to 24 months post-surgery
Failure rate | up to 24 months
  Number of readmission for meniscus tear

SECONDARY OUTCOMES:
Change in integrity of meniscus and adjacent tissues (cartilage, bone, synovial tissue) | 12 months after treatment
  Imaging: MRI
Rate of suture type-associated complications | up to 24 months
  Post-operative data collection: inflammation, pain, recurrent tear of the meniscus, instability or stiffness joint, perimeniscal cyst formation, hemarthrosis or effusion.

CONTACTS AND LOCATIONS:
Overall Officials: Robin MARTIN, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois - CHUV, Lausanne, Canton of Vaud
  - Dr Robin MARTIN, Lausanne, Canton of Vaud